CLINICAL TRIAL: NCT06923007
Title: Study on the Safety and Efficacy of VNS in the Treatment of Mild and Moderate AD Patients; a Multi-center, Randomized, Double-blind, Placebo Parallel Control Trial
Brief Title: Alzheimer's Disease Treated With Vagus Nerve Stimulation
Acronym: Advant
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Municipal Administration of Hospitals (Other Government)
Responsible Party: Principal Investigator, Zhang Jianguo, Director of functional neurosurgery in Beijing Tiantan Hospital, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZLRK202313
Record Dates: First submitted 2025-04-09; First posted 2025-04-11 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Alzheimer Disease (AD)
Keywords: VNS; vagus nerve stimulation
MeSH Terms: conditions — Alzheimer Disease | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, double-blind, placebo, parallel control trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, therapists, care providers, investigators, and outcomes assessors do not know which group (VNS or sham-VNS) the patients are randomized. Only the programmer who programs the device settings knows which group the subject is randomized into.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vague nerve stimulation group (Experimental): Participants receive active vagus nerve stimulation (VNS) for 6 months.
  Interventions: Device: Vagus Nerve Stimulation
- Sham VNS group (Sham Comparator): Participants receive sham vagus nerve stimulation for 6 months.
  Interventions: Device: Sham Vagus Nerve Stimulation

INTERVENTIONS:
Device: Vagus Nerve Stimulation — After randomization, VNS is performed for 6 months. The stimulation parameters will be 30 Hz and 250 μs, the maximum tolerable current is selected according to the patients' adverse reactions (dizziness, palpitations, abnormal sensations, local pain, etc.), and the recommended treatment intensity is 0.8 mA.
  Arms: Vague nerve stimulation group
Device: Sham Vagus Nerve Stimulation — After randomization, sham vagus nerve stimulation VNS treatment is performed for 6 months. The stimulation parameters will be 30 Hz, 250 μs, and the treatment intensity will be 0 mA.
  Arms: Sham VNS group

SUMMARY:
The goal of this clinical trial is to evaluate the safety and efficacy of vagus nerve stimulation (VNS) for treating Alzheimer's disease (AD) in patients aged 50-80 years with mild cognitive impairment to moderate Alzheimer's disease. The main questions it aims to answer are:

Is the change from baseline in the Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog14) score at 6 months post-randomization better in the VNS group compared to the sham stimulation group? Is the change from baseline in scores of other cognitive function, neuropsychiatric symptom, or activities of daily living scales at 6 months post-randomization better in the VNS group compared to the sham stimulation group? Researchers will compare the group receiving vagus nerve stimulation (active VNS group) and the group receiving sham vagus nerve stimulation (sham VNS group) to see if VNS is more effective in improving cognitive function, neuropsychiatric symptoms, or activities of daily living.

Participants will:

Undergo screening assessments (including medical history, physical exams, cognitive and behavioral scale assessments, imaging, etc.).

Undergo surgery for VNS device implantation. Be randomized to either the active VNS or sham VNS group and receive the corresponding stimulation treatment for 6 months (while continuing standard AD medication).

Attend multiple follow-up visits during the study (baseline, randomization day, 3 months, and 6 months post-randomization) for clinical scale assessments.

Potentially provide biological samples (blood, CSF) and undergo additional auxiliary examinations (e.g., MRI, EEG, PET) at specific time points.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 50-80 years
2. Subjects conform to the diagnostic criteria for AD established by the National Institute on Aging and the Alzheimer's Association [National Institution Aging and Alzheimer's Association (NIA-AA)]
3. There is mild to moderate cognitive impairment, and the clinical cognitive rating scale [Clinical Dementia Rating (CDR)] score is 0.5-2.
4. Stable use of the drug for more than 1 month, and no plan to change the medication within 6 months after randomization
5. The informed consent form is signed, and the patient complies with the requirements.

Exclusion Criteria:

1. Dementia caused by other reasons, including vascular dementia, central nervous system infections (such as AIDS, syphilis, etc.), Creutzfeldt-Jakob disease, Huntington's disease and Parkinson's disease, dementia with Lewy bodies, traumatic brain injury dementia, other physical and chemical factors (such as drug poisoning, alcohol poisoning, carbon monoxide poisoning, etc.), significant physical illnesses (such as hepatic encephalopathy, pulmonary encephalopathy, etc.), intracranial space-occupying lesions (such as subdural hematoma, brain tumor), endocrine system disorders (such as thyroid disease, parathyroid disease), and dementia due to vitamin deficiency or any other cause.
2. The presence of a serious or unstable disease, including cardiovascular, liver, kidney, gastrointestinal, respiratory, endocrine, neurological (AD-derived cognitive impairment excluded), psychiatric, immune or blood disorders, and other diseases that the investigator considers may affect the analysis results of this study, or life expectancy < 24 months.
3. A history of cancer within 5 years, except for non-metastatic basal cell carcinoma and/or squamous cell carcinoma, cervical carcinoma in situ, non-progressive prostate cancer, or other cancers with low risk of recurrence or spread.
4. The subject has been diagnosed with any primary mental disorder other than AD-related cognitive impairment. If the investigator deems that the presence of this mental disorder or symptom may affect the interpretation of VNS efficacy, cognitive assessment, or the subject's ability to complete the study, then the subject imust be excluded. Subjects with a history of schizophrenia or other chronic psychiatric conditions are also excluded.
5. Subjects who are judged by the investigator to have suicidal tendencies
6. Illiteracy or insufficient education to complete the scale assessment
7. Having a history of alcohol or drug abuse (excluding smoking history) within 2 years prior to the screening visit
8. A history of multiple or severe drug allergy, obvious atopic allergic constitution or severe hypersensitivity after treatment (including but not limited to severe polymorphic erythema, linear IgA dermatosis, toxic epidermal necrolysis and/or exfoliative dermatitis) with clinical significance
9. Important abnormalities that may be clinically significant and harmful to the subject, affect the study, or suggest other evidence of etiology of dementia during screening, such as physical examination or neurological examination, vital signs, ECG or clinical laboratory test results (determined by the investigator)
10. Screening MRI results showing significant abnormalities suggest another potential cause of progressive cognitive impairment, or findings with clinical significance that may affect the participants ability to safely participate in the study. For example, more than two infarcts larger than 2 cm in diameter, infarcts in critical areas such as the thalamus, hippocampus, internal olfactory cortex, parahippocampal cortex, angular gyrus, or other gray matter nuclei in the subcortical regions, as well as a score of > 2 on the Fazekas Scale
11. Any MRI contraindications, including claustrophobia, or the presence of prohibited metal (ferromagnetic) implant/cardiac pacemakers
12. There are contraindications for VNS surgery, such as left vagus nerve injury, severe infection at the surgical site, and severe heart, lung, liver, kidney or other system dysfunction that cannot tolerate general anesthesia surgery.
13. Currently participating in other interventional clinical trials, or any other type of medical research that is considered scientifically or medically incompatible with this study
14. Other reasons that hinder the completion of this study, such as lack of stable caregivers
15. Female subjects who are pregnant or planning to become pregnant
16. Research center staff members and/or their immediate family members directly related to this study. Immediate family members are spouses, parents, children, or siblings, whether biological or legally adopted relatives.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in ADAS-Cog 14 Score | Baseline, 6 Months Post-randomization
  Change from baseline in the Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) 14-item total score. The ADAS-Cog assesses the severity of cognitive symptoms of Alzheimer's disease. Higher scores indicate greater cognitive impairment. Change is calculated as the score at a given timepoint minus the score at baseline.

SECONDARY OUTCOMES:
Change From Baseline in MMSE Score | Baseline, 6 Months Post-randomization
  Change from baseline in the Mini-Mental State Examination (MMSE) score. Assesses global cognitive function. Scale ranges from 0 to 30; higher scores indicate better cognitive function. Change = Score at Timepoint - Score at Baseline.
Change From Baseline in AVLT Scores | Baseline, 6 Months Post-randomization
  Change from baseline in the Auditory Verbal Learning Test (AVLT) scores. Assesses verbal learning and memory. Key sub-scores assessed include immediate recall (sum of trials 1-5) and delayed recall. Scale ranges from 0 to 84; higher scores indicate better cognitive function.Change = Score at Timepoint - Score at Baseline.
Change From Baseline in CDR-SB Score | Baseline, 6 Months Post-randomization
  Change from baseline in the Clinical Dementia Rating - Sum of Boxes (CDR-SB) score. Assesses dementia severity across 6 domains (Memory, Orientation, Judgment & Problem Solving, Community Affairs, Home & Hobbies, Personal Care). Scores range from 0 to 18; higher scores indicate greater impairment. Change = Score at Timepoint - Score at Baseline.
Change From Baseline in CDR-GS Score | Baseline, 6 Months Post-randomization
  Change from baseline in the Clinical Dementia Rating - Global Score (CDR-GS). Provides an overall dementia severity stage (0=Normal, 0.5=Questionable, 1=Mild, 2=Moderate, 3=Severe) based on cognitive and functional performance. Change = Score at Timepoint - Score at Baseline.
Change From Baseline in HAMA Score | Baseline, 6 Months Post-randomization
  Change from baseline in the Hamilton Rating Scale for Anxiety (HAMA) total score. Assesses the severity of anxiety symptoms across 14 items. Higher scores indicate greater anxiety. Change = Score at Timepoint - Score at Baseline.
Change From Baseline in MAES Score | Baseline, 6 Months Post-randomization
  Change from baseline in the Modified Apathy Evaluation Scale (MAES) score. Assesses the severity of apathy. Higher scores indicate greater apathy. Change = Score at Timepoint - Score at Baseline.
Change From Baseline in ADCS-ADL Score | Baseline, 6 Months Post-randomization
  Change from baseline in the Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) Inventory score. Assesses patient functional ability in activities of daily living based on caregiver report. Higher scores indicate better functional ability. Change = Score at Timepoint - Score at Baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Jianguo Zhang, MD, Principal Investigator — Department of Neurosurgery, Beijing Tiantan Hospital, Capital Medical University, Beijing, China; Wei Zhang, MD, Principal Investigator — Department of Neurology, Beijing Tiantan Hospital, Capital Medical University, Beijing, China
Locations (1):
- Beijing Tiantan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No